CLINICAL TRIAL: NCT05220514
Title: Mayo Clinic Health System-wide Neurological, Vascular and Neurovascular Events With SARS-CoV-2- Part II
Brief Title: Long-term Effects of COVID-19
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Young M. Erben, Principal Investigator, Mayo Clinic
Other Study IDs: 21-008855; R35NS097273 (NIH)
Record Dates: First submitted 2022-01-10; First posted 2022-02-02 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: COVID-19; SAR-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — PK 11195; 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-COVID-19 Diagnosis Control Group: Subjects hospitalized and receiving intensive care for diagnosis of an acute neurological disease other than COVID-19
  Interventions: Drug: (R)-1-(2-chlorophenyl)- N-[11C] ([11C] PK11195); Drug: 2-(4-[11C]methylamino phenyl)-6-hydroxybenzothiazole (11C]6-OH-BTA-1 or [11C]PIB)
- COVID-19 Diagnosis Case Group: Subjects previously hospitalized at Mayo Clinic Hospital for treatment of PCR test confirmed COVID-19
  Interventions: Drug: (R)-1-(2-chlorophenyl)- N-[11C] ([11C] PK11195); Drug: 2-(4-[11C]methylamino phenyl)-6-hydroxybenzothiazole (11C]6-OH-BTA-1 or [11C]PIB)

INTERVENTIONS:
Drug: (R)-1-(2-chlorophenyl)- N-[11C] ([11C] PK11195) — Radiotracer used during the PET-MR scan of the study to identify signs of disease. Used in studies related to Alzheimer's disease. Only FDA approved for investigational use.
Drug: 2-(4-[11C]methylamino phenyl)-6-hydroxybenzothiazole (11C]6-OH-BTA-1 or [11C]PIB) — Radiotracer used during the PET-MR scan of the study to identify signs of disease. Used in studies related to Alzheimer's disease. Only FDA approved for investigational use.

SUMMARY:
The purpose of this study is to measure, monitor, and analyze long term effects of SARS-CoV-2. The main purpose is to assess the post-hospitalization outcomes of patients who were diagnosed with SAR-CoV-2 by comparing to patients who were hospitalized with an acute neurological disease.

ELIGIBILITY:
Inclusion Criteria:

* Control Participants: Males and females over the age of 18 years hospitalized and receiving intensive care for diagnosis's other than COVID-19 or an acute neurological disease and who were not diagnosed (clinically or with PCR testing) with COVID-19.
* Case Participants: Males and females over the age of 18 years who had been hospitalized at Mayo Clinic Hospital for treatment of COVID-19 confirmed by PCR test.
* We acknowledge that some participants may be unable to consent due to underlying medical conditions; an eligible proxy may provide the informed consent and provide a signature on the designated line.
* Women of childbearing age, between the ages of 18 to 55, must complete a negative pregnancy test.
* Minority individuals over the age of 18 years will be eligible to enroll.

Exclusion Criteria:

* Males and females, under the age of 18 years.
* Participants with PET/MRI non-compatible devices.
* Claustrophobia.
* Allergies to study related procedures.
* Pregnant , incarcerated, or institutionalized subjects will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample size of 100 patients hospitalized for COVID-19 with a subset of control patients hospitalized and receiving intensive care for diagnosis other than COVID-19 or an acute neurological disease.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in neurological, cognitive, and functional trajectories in participants who are status post hospitalization for COVID-19 and participants receiving intensive care for diagnosis other than COVID-19 | Baseline, 9 months, 12 months, 24 months.
  Collect participants' self reported response from questionnaire: Post-Covid Functional Status.
Change in neurological, cognitive, and functional trajectories in participants who are status post hospitalization for COVID-19 and participants receiving intensive care for diagnosis other than COVID-19 | Baseline, 9 months, 12 months, 24 months.
  Collect participants' self reported response from questionnaire: Questionnaire for Verifying stroke-free Status.
Change in neurological, cognitive, and functional trajectories in participants who are status post hospitalization for COVID-19 and participants receiving intensive care for diagnosis other than COVID-19 | Baseline, 9 months, 12 months, 24 months.
  Collect participants' self reported response from questionnaire: Patient Health Questionnaire.
Change in neurological, cognitive, and functional trajectories in participants who are status post hospitalization for COVID-19 and participants receiving intensive care for diagnosis other than COVID-19 | Baseline, 9 months, 12 months, 24 months.
  Collect participants' self reported response from questionnaire: Six-Item Screener.
Change in neurological, cognitive, and functional trajectories in participants who are status post hospitalization for COVID-19 and participants receiving intensive care for diagnosis other than COVID-19 | Baseline, 9 months, 12 months, 24 months.
  Collect participants' self reported response from questionnaire: Modified Rankin Scale.
Change in neurological, cognitive, and functional trajectories in participants who are status post hospitalization for COVID-19 and participants receiving intensive care for diagnosis other than COVID-19 | Baseline, 9 months, 12 months, 24 months.
  Collect participants' self reported response from questionnaire: Clinical Dementia Rating.
Change in neurological, cognitive, and functional trajectories in participants who are status post hospitalization for COVID-19 and participants receiving intensive care for diagnosis other than COVID-19 | Baseline, 9 months, 12 months, 24 months.
  Collect participants' self reported response from questionnaire: National Institutes of Health Stroke Scale.
Change in neurological, cognitive, and functional trajectories in participants who are status post hospitalization for COVID-19 and participants receiving intensive care for diagnosis other than COVID-19 | Baseline, 9 months, 12 months, 24 months.
  Collect participants' self reported response from questionnaire: Neuropsychiatric Inventory Questionnaire.
Change in neurological, cognitive, and functional trajectories in participants who are status post hospitalization for COVID-19 and participants receiving intensive care for diagnosis other than COVID-19 | Baseline, 9 months, 12 months, 24 months.
  Collect participants' self reported response from questionnaire: Epworth Sleepiness Scale.
Change in neurological, cognitive, and functional trajectories in participants who are status post hospitalization for COVID-19 and participants receiving intensive care for diagnosis other than COVID-19 | Baseline, 9 months, 12 months, 24 months.
  Collect participants' self reported response from questionnaire: National Alzheimer's Coordinating Center Unified Data Set
Change in neurological, cognitive, and functional trajectories in participants who are status post hospitalization for COVID-19 and participants receiving intensive care for diagnosis other than COVID-19 | Baseline, 9 months, 12 months, 24 months.
  Collect participants' self reported response from questionnaire: Unified Parkinson Disease Rating Scale III.
Change in neurological, cognitive, and functional trajectories in participants who are status post hospitalization for COVID-19 and participants receiving intensive care for diagnosis other than COVID-19 | Baseline, 9 months, 12 months, 24 months.
  Collect participants' self reported response from questionnaire: Montreal Cognitive Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Young Erben, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials